CLINICAL TRIAL: NCT07192224
Title: Effect of Intravenous Fluid Warmer on Prevention of Hypothermia in Laparoscopic Gastrointestinal Cancer Surgeries During General Anesthesia
Brief Title: Efficacy of IV Fluid Warmer for the Prevention of Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-23-03
Record Dates: First submitted 2025-09-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-03

CONDITIONS: Hypothermia; Shivering
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hotline (Experimental): These patients had fluid via hotline.
  Interventions: Device: Hotline
- Placebo (Placebo Comparator): Received fluid at room temperature.
  Interventions: Device: Hypothermia

INTERVENTIONS:
Device: Hypothermia — This study involves the comparison of 2 groups, one receiving warm fluids while the other group receiving room temperature fluids during surgeries.
  Arms: Placebo
Device: Hotline — Used as a fluid warmer.
  Arms: Hotline

SUMMARY:
This study focuses on the importance of the maintenance of body temperature during the surgeries. This study involves the comparison of 2 groups, one receiving warm fluids while the other group receiving room temperature fluids during surgeries.

DETAILED DESCRIPTION:
This study focuses on the importance of the maintenance of body temperature during the surgeries. This study involves the comparison of 2 groups, one receiving warm fluids while the other group receiving room temperature fluids during surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years,
2. ASA I-II,
3. both Male & female,
4. elective gastrointestinal cancer surgery -

Exclusion Criteria:

1. Preoperative core temperature greater than 37.2,
2. severe endocrine respiratory & cardiovascular disease. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
hypothermia | 5-6 months
  Prevention of hypothermia

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanam Memorial Cancer Hospital LAHORE, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
To maintain the confedentiality